CLINICAL TRIAL: NCT02063633
Title: Radiotherapeutic Tumor Response and Normal Tissue Effect in Treating Thoracic Malignancy : as Comparing With Free-breathing Non-gating Methods.
Brief Title: PET With Respiratory Gating Technique in Evaluation of Response and Normal Tissue Effect in Thoracic Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102118-F
Record Dates: First submitted 2014-02-07; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: To Correlate RPM Respiratory-gating Methods Analyses, Treatment Response, and Normal Tissue Metabolic Effect.; Application in Clinical Outcomes and Prediction of Prognosis.
Keywords: Thoracic malignancy, irradiation, respiratory gating system PET

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Technologic advances in the field of radiation oncology have made in possible to deliver a highly conformal and accurate radiation dose to a target tissue. Accompanying the rapid implementation of these novel techniques is often a reduction in the radiation margins, which reinforces the importance of accurate target delineation, and reduces the side effect of therapy.

F-18 FDG PET/CT is widely used in oncology, including complete whole body staging, restaging and monitoring of tumor response in different types of cancers. As to non-oncology application, inflammation in almost any tissue will result in increased FDG accumulation. However, the normal tissue with sparing radiation may show subtle change, and would be difficult to be detected. FDG PET/CT was limited in the spatial resolution of 5 mm and low FDG-avid disease. To be evaluation of the interval change of metabolic response before and after radiotherapy of thoracic malignancies, we plan to initiate a prospective study trail the takes advantages of recent technical advances of technique in 4-dimensional PET/CT (4-D PET/CT) with respiratory gating system.

Respiratory motion creates artifacts in PET and PET/CT images, and can alter diagnosis. The tumor edge would be blurred due to respiratory movement, and be underestimated the uptake value. Also, semi-quantitative measurement, standard uptake value (SUV), combined with parameters such as the lesion site and shape, which is commonly used to make the final assessment of disease would be mis-estimated.

The study aims to investigate the correlation of 4-D PET/CT with respiratory gating methods and free breathing PET/CT when processing primary thoracic malignancy and normal tissue effect.

DETAILED DESCRIPTION:
Radiation pneumonitis is the dose-limiting toxicity in thoracic radiotherapy (RT) for thoracic malignancy. It occurs beginning after the initiation of RT for up to 6 months characterized by cough, shortness of breath, and changes in lung function. A mortality rate approaches 50% in severe radiation pneumonitis [4]. Dosimetric parameters, such as the percentage of lung volume irradiated ≧20 Gy (V20) and the mean lung dose (MLD), provide a guide to assess the risk of radiation pneumonitis in the treatment planning process. However, the parameters have poor predictive power for individual risk. The appearance of radiation lung injury shown in computed tomography (CT) was characterized by and early and a late phase. Since, radiation pneumonitis is characterized by the migration of leukocytes from the blood to irradiated lung tissue; thus, on FDG-PET imaging, more intense inflammatory responses will result in greater FDG uptake. Identifying an early sign or precursor of normal tissue damage helps predicting the delayed organ dysfunction.

In combined PET/CT, CT is used for localization and correction for attenuation in the PET images. An accurate spatial registration of PET and CT image sets is a prerequisite for accurate diagnosis and SUV measurement. However, because of respiration, and the difference in the acquisition time required to image the thorax between PET (6-9 minutes) and CT (~15 seconds), spatial misalignment between the 2 image sets is not uncommon. This misalignment significantly compromises the interpretation of PET images, resulting in mislocalization of the lesion and inaccurate quantitation of the SUV. The main cause of these artifacts is the dynamic interaction between transaxial image acquisition and the asynchronous motion of tumor and normal tissues. To account for motion effects, respiratory gating techniques have been developed.

A more sophisticated respiratory-motion monitoring system is the Real-Time Position Management respiratory gating system (RPM). The system includes a video camera that measures respiratory motion by tracking the vertical displacement of 2 infrared reflective markers rigidly mounted on a plastic block placed on the patient's thorax. The motion of the block is displayed by a graphical interface on the RPM workstation. It has been used in gated radiotherapy of lung, respiratory-gated CT, and 4-D CT, as well as respiratory-gated PET imaging.

We plan to enroll patients with thoracic cancer who scheduled further radiotherapy. Patients with pre-existing chronic lung disease, such as COPD, interstitial lung disease, cystic lung disease, et al, will be excluded. The FDG PET/CT will be performed before the radiotherapy (baseline study), and 30-45 days after completing radiotherapy (2nd study). Free-breathing whole body scan will be performed after 40 minutes, and regional 4D PET/CT with RPM method for chest was performed subsequently. These patients will be follow-up in radiation oncology clinics, any radiation-related adverse effect and long-term prognosis will be recorded. The association between the data analysis will be further investigated.

We will obtain better delineation of the correlation and the differences between free-breathing PET/CT 4-D PET/CT with RPM respiratory-gating methods in processing tumor metabolism, more over, to assess normal tissue metabolic effect. And the further work is trying to find if the application helps in clinical outcomes and prediction of prognosis of the technique of 4-D PET/CT with RPM respiratory-gating methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thoracic cancer who will be scheduled further radiotherapy.
* Aged 20-80 years old.

Exclusion Criteria:

* Pre-existing chronic lung disease, such as COPD, interstitial lung disease, cystic lung disease, et al.
* Pregnancy.
* Any medical contraindication of FDG PET study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thoracic cancer who will be scheduled further radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
normal tissue effect | Dec, 2014
  The patient should be fasting prior to the exam for at least 6 hours. Before the radiopharmaceutical injection, we will take a sample of blood from a vein to test the blood sugar level. High levels of circulating glucose essentially compete with radioactive FDG in the exam, and image degradation may occur. Then F-18 FDG PET/CT study with 10 mCi tracer was injected from vein. All PET/CT studies were performed on the hybrid PET/CT scanner (Discovery VCT, General Electric Medical Systems).After uptake time of 60 minutes, whole body FDG PET from the vertex of the skull to the proximal thighs in 3D mode at 60 minutes after intravenous administration of FDG. After 60 minutes of the first imaging, delayed 4-D PET/CT with RPM respiratory gating method will be applied to lung fields. The time-points of FDG PET/CT are before radiotherapy (baseline study), and 30-45 days after completing radiotherapy (2nd study).

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan